CLINICAL TRIAL: NCT00678678
Title: Chest Physiotherapy After Bariatric Surgery - a Comparison Between Incentive Spirometry and Epap
Brief Title: Chest Physiotherapy After Bariatric Aurgery - A Comparison Between Incentive Spirometry and Expiratory Positive Airway Pressure (Epap)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Other Study IDs: 01/07
Record Dates: First submitted 2008-04-29; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
Keywords: Physiotherapy; Breathing exercises; Bariatric Surgery; Laparoscopy
MeSH Terms: conditions — Obesity

ARMS (2):
- I - Spirometer (Active Comparator)
  Interventions: Device: Incentive Spirometry - RESPIRON
- II - Kit Epap® (Active Comparator): Device with Spring load by mask,produced by Brazil (critical med)
  Interventions: Device: Kit Epap®:

INTERVENTIONS:
Device: Incentive Spirometry - RESPIRON — Device that stimulates the deep breathing, flow-oriented
  Arms: I - Spirometer
Device: Kit Epap®: — Device that providing constant positive pressure during expiration, given by spring load (cmH2O), using a face mask as an interface
  Other Names: EPAP - End positive airway pressure; Spring Load by mask
  Arms: II - Kit Epap®

SUMMARY:
Objective: To compare the effects of the EPAP and the incentive spirometry flow-oriented in the pulmonary function after bariatric surgery.

Method: Twenty-eight women, non-smokers, with no lung disease and BMI of 35-49,99 kg/m2, undergoing bariatric surgery by laparoscopy, were studied. Before surgery the patients were divided in two groups: Spirometer Group (SG) (n=13) and EPAP Group (EG) (n=15). Pulmonary function was evaluated by spirometry, thoracoabdominal (cirtometry) and diaphragmatic motion, on the preoperative and on the second postoperative day. Physiotherapy started on the day of surgery, each modality (incentive spirometry or EPAP) performed lasting 15 minutes. The deambulation and active exercises of upper and lower limbs were standardized for groups.

ELIGIBILITY:
Inclusion Criteria:

* Obese with body mass index between: 35 e 50 kg/m2
* Non-smokers
* No lung disease

Exclusion Criteria:

* Unable to perform the evaluation tests
* Not signed the consentment term

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
spirometry, thoracoabdominal (cirtometry) and diaphragmatic motion | preoperative and second postoperative day

SECONDARY OUTCOMES:
Hospital stay and postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Meridional Hospital, Cariacica, Espírito Santo, Brazil